CLINICAL TRIAL: NCT05836558
Title: Are the Results of Minimally Invasive Mitral Valve Repair Still Satisfactory When Looked at Very Long-term
Brief Title: Are the Results of Minimally Invasive Mitral Valve Repair Still Satisfactory When Looked at Very Long-term?
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: VLTFUP-MINIMVR
Record Dates: First submitted 2023-01-27; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mitral valve repair in right minithoracotomy — reparative surgery of the mitral valve accessing heart via an incision in the right 3rd or 4th intercostal space.

SUMMARY:
Mitral regurgitation (MR) is a disease affecting the mitral valve that it causes a volumetric and pressure overload in the left chambers due to the leak of the unidirectionality normally guaranteed by the heart valve system.

The gold standard for severe mitral regurgitation is currently surgical mitral valve repair (PLM) using longitudinal median sternotomy to expose the heart Since the mid-1990s, the right mini-thoracotomy, ie a surgical access with cut in the 3rd or 4th intercostal space that would allow to reduce the size of the surgical site making it less traumatic and more aesthetic, addressing mainly a young target population.

Since the 2000s this method has spread more and more, expanding all over the world and spreading especially in the United States and Germany. This method has been progressively used in the treatment of the whole mitral valve surgery starting from valve repair up to prosthetic replacements.

Mitral valve repair through minimally invasive access in degenerative pathology has made it possible to obtain excellent long-term results, with low recurrence rates of regurgitation. In our center the results on the first 48 patients have been published in 2005 by Lapenna et al. Over the years this method has been adopted in thousands of patients worldwide, however the data present in the literature they stop at a follow-up of about 10 years. In 2017 De Bonis et al. of the San Raffaele Hospital have published the outcome of a particular subgroup of patients (bileaflet prolapse) treated with minimally invasive access, comparing them with as many subjects subjected to the same method of mitral repair ("edge-to-edge technique or Alfieri stitch"), obtaining superimposable long-term results (about 14 years old).

The goal of the present study is to analyze very long-lasting results in patients treated with mitral valve surgery with access in right mini-thoractotomy.

ELIGIBILITY:
Inclusion Criteria:

* patients with degenerative mitral regurgitation
* patients treated with mitral valve repair in right minithoracotomy

Exclusion Criteria:

* median sternotomy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients operated with mitral valve repair in right minithoracotomy to treat degenerative mitral valve disease
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, a minimum of 16 years

SECONDARY OUTCOMES:
Reintervention | through study completion, a minimum of 16 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided